CLINICAL TRIAL: NCT03975621
Title: Nurse AMIE: A Tablet Based Supportive Care Platform in Metastatic Breast Cancer (AMIE = Addressing Metastatic Individuals Everyday)
Brief Title: Nurse AMIE: Addressing Metastatic Individuals Everyday
Acronym: NurseAMIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Kathryn Schmitz, Professor, Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00011444
Record Dates: First submitted 2019-06-04; First posted 2019-06-05 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Metastatic Breast Cancer
Keywords: Exercise; Feasibility; Acceptability; Supportive Care Platform
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention (Experimental): The immediate intervention group will receive the intervention at the time of consent (baseline) and will be enrolled in the intervention for a total of 6 months. Patients will receive the tablet, a pedometer and an exercise band. Patients will use Nurse AMIE while receiving weekly phone calls from a patient navigator. After 90 days of the intervention observation will take place for 90 days, the patient will be asked to continue using Nurse AMIE without a patient navigator's presence.
  Interventions: Behavioral: Supportive Care
- Delayed Intervention (Experimental): The delayed intervention group will receive the intervention 3 months after consent (6 months of intervention with 3 months delay total of 9 months); the patient will then follow the same pattern as listed above. The only difference is we will ask the delayed intervention group to wear a FitBit device for 1 week following consent in order to gain baseline data as to their activity/movement.
  Interventions: Behavioral: Supportive Care

INTERVENTIONS:
Behavioral: Supportive Care — Patient will receive the tablet, a pedometer (to track their steps) and an exercise band (to complete the exercise videos). Use of Nurse AMIE while receiving intervention phone calls from a patient navigator.
  After 90 days, observation begins and the patient will be asked to continue using Nurse AMIE without a patient navigator's presence.

SUMMARY:
Determine the acceptability and feasibility of a supportive care software platform to improve quality of life and function in metastatic breast cancer patients. Acceptability will be defined as the proportion of women offered the intervention who agree to participate. Feasibility will be defined as the proportion of women who consent, take a tablet home, who actually interact with the tablet and participate at least one month of the program.

DETAILED DESCRIPTION:
Goals of the Nurse AMIE software program are to regularly assess psychosocial, functional, and symptom needs among metastatic breast cancer patients and to provide appropriate interventions via YouTube style videos, weekly phone calls with a patient navigator at Penn State, and appropriate referrals to phone or in person consultations as needed. The proposed Nurse AMIE software program will allow for the provision of resources (YouTube style videos, audio files, exercises) to intervene on many of the common symptoms and challenges experienced by metastatic patients. This is an identified need on the part of both metastatic patients and their medical care teams. Finally, it will also allow patient navigators to check in with patients, reviewing responses to surveys, discerning whether new or different interventions are needed, and connecting women to palliative care and other services if additional care is warranted.

ELIGIBILITY:
Inclusion Criteria:

* Women with metastatic breast cancer
* ECOG performance score ≤3.
* English Speaking
* With sufficient vision/hearing or family support
* Willingness to be randomized

Exclusion Criteria:

* Medical or psychiatric conditions (beyond breast cancer, its treatment, and its symptoms) that would impair our ability to test study hypotheses (e. g. psychotic disorders, dementia, inability to give informed consent or follow the instruction).
* Patients who are receiving any other behavioral intervention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of the Application: The proportion of women who consent, take a tablet home, who actually interact with the tablet and participate at least one month of the program. | 3 Months
  Feasibility is defined as the proportion of women who consent, take a tablet home, who actually interact with the tablet and participate at least one month of the program.

SECONDARY OUTCOMES:
Acceptability of the Application: The proportion of patients who agree to participate among those deemed eligible and cleared by oncologist. | 3 Months
  The proportion of patients who agree to participate among those deemed eligible and cleared by oncologist.

OTHER OUTCOMES:
Quality of Life: Short Form 36 | Through study completion, an average of 9 months
  The Short Form 36 Health Survey (SF-36) is a 36-item, patient-reported survey of patient health. The SF-36 is a measure of health status and an abbreviated variant of it.
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Quality of Life: Functional Assessment of Cancer Therapy- Breast | Through study completion, an average of 9 months
  The Functional Assessment of Cancer Therapy-Breast (FACT-B), is a 44-item self-report instrument designed to measure multidimensional quality of life (QOL) in patients with breast cancer.
  The FACT-B questionnaire includes 44 items, consisting of 5 subscales, all subscale items are summed to a total. The higher the score the better QOL
Physical Function: Short Physical Performance Battery | Through study completion, an average of 9 months
  Objectively-measured physical function will be assessed using the Short Physical Performance Battery (SPPB). The SPPB is an accumulation of balance tests, 4-meter gait speed, and 5-chair stands. Based on the time needed to complete the chair stands, a score is given. A summation of scores from all tests is taken, ranging from 0 -12. A higher score = Higher physical function.
Sleep: Sleep Quality Assessment (PSQI) | Through study completion, an average of 9 months
  Sleep quality and sleep problems will be assessed with the validated and frequently used Pittsburgh Sleep Quality Index (PSQI).
  In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Pain: Brief Pain Inventory (Short Form) | Through study completion, an average of 9 months
  Bodily pain will be assessed using the Brief Pain Inventory- Short form (BPI-SF).
  The BPI gives two main scores: a pain severity score and a pain interference score. The pain severity score is calculated from the four items about pain intensity. Each item is rated from 0, no pain, to 10, pain as bad as you can imagine, and contributes with the same weight to the final score, ranging from 0 to 40. The pain interference score corresponds to the item on pain interference. The seven sub-items are rated from 0, does not interfere, to 10, completely interferes, and contributes with the same weight to the final score, ranging from 0 to 70.
Fatigue: Brief Fatigue Inventory | Through study completion, an average of 9 months
  The Brief Fatigue Inventory (BFI) is used to rapidly assess the severity and impact of cancer-related fatigue. An increasing focus on cancer-related fatigue emphasized the need for sensitive tools to assess this most frequently reported symptom. The six interference items correlate with standard quality-of-life measures.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn H Schmitz, PhD, Principal Investigator — Penn State University
Locations (1):
- Penn State Cancer Institute, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No